CLINICAL TRIAL: NCT00123032
Title: Bright Start: Obesity Prevention in American Indian Children
Brief Title: School- and Home-Based Program to Prevent Obesity in American Indian Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 228
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): This group will focus on improving their diet and increasing physical activity at home and at school.
  Interventions: Behavioral: Diet; Procedure: Exercise
- 2 (No Intervention): A control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Diet — Increase the availability of fruits and vegetables, serve recommended portion sizes and reduce availability of excessive energy-dense foods at school cafeterias to improve the diet of participants at school breakfast, lunch and snacks.
  Arms: 1
Procedure: Exercise — Increase active recess time, implement classroom action breaks and increase school PE class time to increase physical activity among participants.
  Arms: 1

SUMMARY:
The purpose of this study is to prevent excessive weight gain among kindergarten and first grade American Indian children using improved diet and increased physical activity at home and at school.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity has reached epidemic proportions nationwide among children, adolescents, and adults and is considered one of the most serious health problems facing Americans today. There is a higher prevalence of obesity among ethnic minority groups and those with a lower family income. American Indian children and adults are among those with the highest rates of obesity and related diseases. Young American Indians have high rates of type 2 diabetes, and the rates appear to be increasing substantially. Obesity in American Indian children has serious implications for their immediate and long-term health. Unless this trend is reversed, American Indian populations will be burdened by an unprecedented increase in the incidence of chronic diseases, such as type 2 diabetes and cardiovascular disease.

The high prevalence of obesity among American Indian children and the associated health and financial burdens warrant strong and effective prevention efforts. While the prevention of childhood obesity has risen to the top of the list of public health priorities, relatively little research has focused on childhood obesity prevention, especially for high-risk populations. The development and evaluation of innovative, culturally appropriate, and effective strategies to prevent excessive weight gain is critical, particularly for American Indian youth. Early prevention efforts are especially important given the substantial evidence that eating and physical activity habits are established in early childhood and continue into adulthood. Adopting healthy eating and physical activity habits early in life is an effective way of preventing obesity and related diseases. The best intervention to prevent obesity in children should target the two most prominent influences on the young child's eating and physical activity behaviors: the school and the family. Obesity in American Indian children begins very early in life, which suggests that interventions need to begin early. Research has shown that 43% of American Indian 5-6 year olds in South Dakota are already overweight. Thus, targeting children in this young age group may be advantageous.

DESIGN NARRATIVE:

The study involves 14 schools on the Pine Ridge and Rosebud reservations, which are two Lakota reservations in South Dakota. Seven schools will be randomly assigned to the intervention condition and 7 schools to the control condition. Schools will be assigned to one of the two groups after baseline measures have been completed. The focus of this intervention, the Ohiyu lyojanjan - Bright Start Program, is to create dietary and physical activity environmental change at school and home. The intervention will follow 500 children in kindergarten for 16 months through the end of 1st grade. There will be 4 schools on the Rosebud reservation and 10 schools on the Pine Ridge reservation assigned to two groups. The two groups will begin the study one year apart; the first group will have baseline measures assessed in the fall of 2005 and begin the intervention in January 2006, and the second group will have baseline measures assessed in the fall of 2006 and begin the intervention in January 2007. This staggered design will allow for more contact with participating schools and families by key study staff, increased monitoring and control of the intervention within schools, and decreased staff costs. The intervention will focus on changing the school and home environments related to physical activity and food. The school physical activity environmental intervention component will incorporate 60 minutes of daily physical activity at school for kindergarten and 1st grade students through a combination of physical education classes, a classroom walking program, in-class activity breaks, and active morning and afternoon recess. The school food environment intervention will focus on improving school meals (breakfast and lunch), classroom snacks, and teacher classroom food practices. The intervention will target the school food service to decrease availability of high-fat and high-sugar foods, regulate portion control of foods served, and increase fruits (not juice) and vegetables served. The family intervention will address the household food and physical activity environment and family dietary and physical activity behaviors. Because parents of kindergarten children in the selected schools will be recruited for participation prior to the school treatment assignments, it may be problematic to engage all parents without providing anything to those who are assigned to the control condition. To foster parent interest in study participation, parents in the control group will be mailed monthly newsletters with general family recommendations for prevention of excess weight gain.

The major hypothesis is that by the end of the 16-month study, children in the intervention schools will have significantly lower body mass index (BMI) and body fat percentage after adjustment for baseline values, as compared to children in the control schools. The primary outcome measures in children are BMI and percent body fat. Secondary measures include child's total daily physical activity, nutrient and food-group analysis of school meals and snacks, and assessment of classroom food and physical activity practices. Child measures will occur at the beginning of kindergarten, at the end of kindergarten (BMI only), and at the end of the 1st grade. Parents will be surveyed at the beginning of their child's kindergarten year, and when their child is at the end of 1st grade. Parent assessments will include measures of household food availability and reports of their own and their child's eating and physical activity behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in kindergarten at one of the participating elementary schools on the Pine Ridge or Rosebud reservations in South Dakota

Exclusion Criteria:

* Schools who do not meet the criteria stated above and are not willing to sign the memorandum of agreement outlining expectations of the school and the University of Minnesota.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
BMI of children | Fall 2005 through Summer 2008
Percentage of body fat of children (measured at the end of the 1st grade school year) | Baseline and followup

SECONDARY OUTCOMES:
Total daily physical activity level of children | Daily during intervention period
Nutrient and food group analysis of school meals and snacks | Baseline and followup
Assessment of classroom food and physical activity practices | Daily during intervention period
Measures of household food availability | Baseline and followup
Parent reports of their eating and physical activity behaviors | Baseline and followup
Parent reports of their children's eating and physical activity behaviors (measured at the end of the 1st grade school year) | Baseline and followup

CONTACTS AND LOCATIONS:
Overall Officials: Mary Story, MD, Study Chair — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Twin Cities, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Zhang J, Himes JH, Hannan PJ, Arcan C, Smyth M, Rock BH, Story M. Summer effects on body mass index (BMI) gain and growth patterns of American Indian children from kindergarten to first grade: a prospective study. BMC Public Health. 2011 Dec 23;11:951. doi: 10.1186/1471-2458-11-951. PMID 22192795